CLINICAL TRIAL: NCT00653250
Title: COX-2 Activity in Early and Advanced NSCLC and The Effect of Short-Term Administration of Specific COX-2 Inhibitors (Celecoxib)
Brief Title: Celecoxib in Treating Patients With Stage I, Stage II, or Stage IIIA Non-Small Cell Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Vicki Keedy, MD, Assistant Professor of Medicine, Medical Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC THO 0055; P50CA090949 (NIH); P30CA068485 (NIH); VU-VICC-THO-0055; VU-VICC-000724
Record Dates: First submitted 2008-04-03; First posted 2008-04-04 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Celecoxib; Biopsy; Transurethral Resection of Bladder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Therapeutic Intervention (Experimental): Correlative
  Interventions: Drug: celecoxib; Procedure: biopsy; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Drug: celecoxib — 400 mg P.O. BID for five days prior to obtaining second serum/urine collection (starting after initial biopsy, serum and urine collection)
  Other Names: celebrex
Procedure: biopsy — in patients with newly diagnosed NSCLC, a pretreatment excision of a small amount of tumor tissue
Procedure: therapeutic conventional surgery — surgery to remove the lung tumor
  Other Names: tumor resection

SUMMARY:
RATIONALE: Studying samples of tissue, blood, and urine from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This clinical trial is studying celecoxib in treating patients with stage I, stage II, or stage IIIA non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess cyclo-oxygenase-2 (COX-2) activity in patients with early-stage non-small cell lung cancer (NSCLC) and correlate the results with serum vascular endothelial growth factor (VEGF) levels, tumor microvessel density score, tumor prostaglandin E2 (PGE_2) and matrix metalloproteinases (MMP) levels, and the major urinary metabolite of PGE_2, PGE-M.
* To assess the effect of specific COX-2 inhibitors (celecoxib) on COX-2 expression within the primary tumor, serum VEGF levels and tumor microvascular density, tumor PGE_2 and MMP levels, and urinary PGE-M in a cohort of patients with early-stage NSCLC.

OUTLINE: Patients receive oral celecoxib 400 mg twice a day for 5 days in the absence of disease progression or unaccepted toxicity. Patients with early-stage disease then undergo surgery.

Biopsy, serum, and urine samples are obtained at baseline and after celecoxib treatment. The biopsy specimen are examined for the expression of cyclo-oxygenase-2 (COX-2), PGE_2, and selected MMPs by immunohistochemistry, western blotting, and northern blotting. Serum and urine samples are analyzed for VEGF and PGE-M expression. COX-2 tumor expression is correlated with serum VEGF levels; tumor MMP-2, MMP-9, and PGE_2 expression; urinary PGE-M and microvessel density scores.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Presumed histological or cytological diagnosis of non-small cell lung cancer

  * Diagnosis to be confirmed upon study entry to collect biopsy material for correlative studies
* Stage I-IIIA disease

PATIENT CHARACTERISTICS:

* ECOG performance status of 0-2
* Serum creatinine ≤ 1.5 mg/dL
* Granulocytes ≥ 1,500/mm^3
* Platelets ≥ 100,000/mm^3
* AST ≤ 3 times normal
* Bilirubin ≤ 1.5 mg/dL
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No active unresolved infection

PRIOR CONCURRENT THERAPY:

* At least 7 days since prior and no concurrent non-steroidal anti-inflammatory agents or other cyclo-oxygenase-2 inhibitors
* At least 7 days since prior parenteral antibiotics
* No prior systemic chemotherapy or radiotherapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2000-12; Primary Completion 2006-03 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Correlation of expression of cyclo-oxygenase-2 (COX-2) activity with serum VEGF levels, tumor microvessel density score, tumor PEG2 and MMP levels, and urinary PGE-M | Date of pretreatment biopsy surgery (tissue) and day 1 (blood)
  COX-2 will be measured in pre-treatment tumor biopsy tissue as well as tumor microvessel density, MMP-2 and PGE2. VEGF will be measured in pre-treatment blood.

SECONDARY OUTCOMES:
Effect of Celecoxib on COX-2 expression and microvascular density in tumor, PGE2 and MMP levels in tumor, serum VEGF levels and urinary PGE-M | After day 5 of 5 days of treatment
  Patients with early-stage NSCLC will undergo tumor resection after 5 days of treatment with celecoxib. Tumor tissue will be examined. Post-treatment blood and urine will also be collected and examined.

CONTACTS AND LOCATIONS:
Overall Officials: Vicki Keedy, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center